CLINICAL TRIAL: NCT03238547
Title: Accuracy of a Semi-quantitative Urine Albumin-to-creatinine Ratio Test as a Screening Tool for Microalbuminuria in Patients With Diabetes
Brief Title: Screening of Microalbuminuria Using a Semi-quantitative UACR Test
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ki Kim, Prof., Seoul National University Hospital
Other Study IDs: URiSCAN_SNU_01
Record Dates: First submitted 2017-07-29; First posted 2017-08-03 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-01

CONDITIONS: Diabetes; Microalbuminuria
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- diabetes: Diabetes patients with normal renal function and normal urinalysis
  Interventions: Diagnostic Test: semi-quantitative urine albumin-to-creatinine ratio test; Diagnostic Test: standard quantitative spot urine albumin-to-creatinine ratio

INTERVENTIONS:
Diagnostic Test: semi-quantitative urine albumin-to-creatinine ratio test — measurement of urine albumin-to-creatinine ratio using URiSCAN 2ACR, a semi-quantitative urine albumin-to-creatinine ratio test
Diagnostic Test: standard quantitative spot urine albumin-to-creatinine ratio — measurement of urine albumin-to-creatinine ratio using a standard turbidimetric immunoassay

SUMMARY:
Microalbuminuria is an important biomarker for the development of diabetic nephropathy and cardiovascular complications. Since microalbuminuria is not easily detected on routine urinalysis, current guidelines recommend measuring spot urine albumin-to-creatinine ratio (uACR) annually in a patient with diabetes mellitus. While the standard method is quantitative measurement using turbidimetric immunoassay, it requires high cost and special laboratory equipment. This may be a hurdle that prevents screening for microalbuminuria in many patients with diabetes. Therefore, a semi-quantitative uACR test, which is rapid and inexpensive, could be used as a substitute to the current standard quantitative measurement. The investigators aimed to assess the diagnostic accuracy of a semi-quantitative urine albumin-to-creatinine ratio test, URiSCAN 2ACR, as a screening tool for microalbuminuria in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* diabetes

Exclusion Criteria:

* microscopic hematuria
* pyuria
* urinary cast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients following Seoul National University Hospital
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic Sensitivity and Specificity | through study completion, an average of 18 months
  Diagnostic Sensitivity and Specificity of URiSCAN 2ACR compared with standard method

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No